CLINICAL TRIAL: NCT06968273
Title: Analysis of Muscle Oxygen Saturation and Functional Variables During Physical Capacity Assessments in Patients With COPD Undergoing a Cardiovascular and Strength Training Program
Brief Title: Analysis of Muscle Oxygen Saturation and Functional Variables During Physical Capacity Assessments in Patients With COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Investigator, University of Extremadura
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 020525
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Muscle Oxygenation; Exercise; Respiratory Physiotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will undergo a 4-week combined respiratory physiotherapy and strength-cardio training program, supervised in hospital. Muscle oxygen saturation and functional variables will be measured pre- and post-intervention.
  Interventions: Behavioral: Combined respiratory physiotherapy and cardiovascular-strength training program

INTERVENTIONS:
Behavioral: Combined respiratory physiotherapy and cardiovascular-strength training program — 20-session supervised hospital-based program including respiratory physiotherapy, aerobic training (guided by Borg scale and HR monitoring), and strength training using progressive loads (based on 1RM). Duration: 4 weeks (5 sessions/week).

SUMMARY:
This experimental pre-post intervention study aims to evaluate the effect of a respiratory physiotherapy and combined strength and cardiovascular training program on muscle oxygen saturation and functional capacity in patients with Chronic Obstructive Pulmonary Disease (COPD). Oxygenation of the intercostal, quadriceps, and triceps surae muscles will be assessed using near-infrared spectroscopy (NIRS) during standard physical performance tests (6-Minute Walk Test and 30-Second Chair Stand Test). Additional functional parameters and quality of life will be recorded pre- and post-intervention. The results will contribute to optimizing rehabilitation programs and monitoring intensity and progress through muscle oxygenation data.

DETAILED DESCRIPTION:
This experimental pre-post study investigates the effects of a combined respiratory physiotherapy and physical training program on muscle oxygen saturation and functional capacity in patients diagnosed with Chronic Obstructive Pulmonary Disease (COPD). COPD is a highly prevalent condition with a progressive impact on functional capacity, muscle performance, and quality of life. It is associated with systemic repercussions, including skeletal muscle dysfunction and oxygen transport limitations, which impair tolerance to physical activity.

The study will evaluate the acute and cumulative effects of a structured, supervised intervention including respiratory physiotherapy techniques, cardiovascular training, and progressive resistance training. Measurements will be taken before and after the intervention period to assess changes in muscle oxygen saturation-measured using near-infrared spectroscopy (NIRS) devices (Moxy Monitor)-in key muscle groups (intercostal, quadriceps, and triceps surae).

Functional capacity will be assessed using the 6-Minute Walk Test (6MWT) and the 30-Second Chair Stand Test (30CST). Additional variables including inspiratory and expiratory pressures, pulmonary function (FEV1/FEV6), heart rate variability, dyspnea, lower limb fatigue, and quality of life (COPD Assessment Test) will also be recorded.

The intervention consists of 20 hospital-based sessions over four weeks (five sessions per week). The protocol is designed to reflect real clinical settings and aims to provide evidence for the feasibility, safety, and functional relevance of combining respiratory and musculoskeletal rehabilitation strategies in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of COPD
* Medically cleared for physical exercise

Exclusion Criteria:

* Decompensated heart failure or exercise-limiting comorbidities
* Cognitive impairment or legal incapacity to consent
* Inability to perform physical tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in muscle oxygen saturation (%) | From baseline to end of intervention (4 weeks)
  Measured in intercostal, quadriceps, and triceps surae muscles using NIRS (Moxy Monitor) during 6MWT and 30CST, before and after the 4-week intervention.

SECONDARY OUTCOMES:
Distance covered in 6-Minute Walk Test (6MWT) | From baseline to after the 4-week intervention
Number of repetitions in the 30-Second Chair Stand Test | From baseline to after the 4-week intervention
Perceived dyspnea and lower limb fatigue (Borg Scale) | From baseline to after the 4-week intervention
Maximal inspiratory and expiratory pressures (Pimax and Pemax) | From baseline to after the 4-week intervention
FEV1/FEV6 ratio (portable COPD Vitalograph) | From baseline to after the 4-week intervention
Heart rate variability and max/min heart rate (Polar system + Kubios HRV) | From baseline to after the 4-week intervention
Quality of life (COPD Assessment Test - CAT) | From baseline to after the 4-week intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saúde do Alto Alentejo (ULSAALE), Hospitals of Portalegre and Elvas, Portugal, Portalegre, Portugal